CLINICAL TRIAL: NCT00667953
Title: Phase I/II Study of Temozolomide and Gleevec (Imatinib Mesylate, Formerly Known as STI571) in Advanced Melanoma
Brief Title: Study of Temzolomide and Gleevec in Advanced Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Difficulty enrolling subjects
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 02602
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Melanoma; Advanced Melanoma
Keywords: Temzolomide; Gleevec; Melanoma; Advanced melanoma; Phase II
MeSH Terms: conditions — Melanoma | interventions — Imatinib Mesylate; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A: (Experimental): Temozolomide plus imatinib
  Interventions: Drug: Gleevec; Drug: Temodar

INTERVENTIONS:
Drug: Gleevec — Gleevec (600 mg) daily.
  Other Names: Imatinib mesylate
Drug: Temodar — Temzolomide (1000 mg/m2) over 5 days on a 28 day cycle.
  Other Names: temozolomide

SUMMARY:
This study has been designed to evaluate the side effects of Gleevec when given in combination with Temzolomide; and to learn more about how these drugs work in the body and whether this combination is useful in treating patients with melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Prior chemotherapy, immunotherapy, radiation therapy (Phase I portion only), cytokine, biologic, or vaccine therapy is permitted, however no prior treatment with temozolomide
* Measurable disease
* Performance status <= 2
* Life expectancy greater than 3 months

Exclusion Criteria:

* No prior treatment with temozolomide or imatinib mesylate
* Organ allografts
* Prior radiotherapy, or prior intratumor injection therapy, to areas of measurable disease that are used as target indicator lesions, unless progression has occurred at that site or measurable disease has developed outside the treatment area
* Pregnancy or lactation
* History of second cancer
* Known hypersensitivity to temozolomide or imatinib
* Use of any experimental therapy within 3 weeks prior to baseline evaluations done prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-01; Primary Completion 2011-03-09 (Actual); Study Completion 2011-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Fecher, MD, Principal Investigator — Rogel Cancer Center; tara mitchell, MD, Study Director — Abramson CC
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Bajor DL, Xu X, Torigian DA, Mick R, Garcia LR, Richman LP, Desmarais C, Nathanson KL, Schuchter LM, Kalos M, Vonderheide RH. Immune activation and a 9-year ongoing complete remission following CD40 antibody therapy and metastasectomy in a patient with metastatic melanoma. Cancer Immunol Res. 2014 Nov;2(11):1051-8. doi: 10.1158/2326-6066.CIR-14-0154. Epub 2014 Sep 24. PMID 25252722

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A:: Gleevec + Temozolomide: Temzolomide (1000 mg/m2) over 5 days on a 28 day cycle. Gleevec (600 mg) daily.
Period: Overall Study
Arm/Group | Arm A:
Started | 32
Completed | 28
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Arm A:
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Safety - Grade 3 or 4 Adverse Events
Description: Number of reported grade 3 or 4 adverse events
Time Frame: through study completion, an average of 1 year
Population: Data from final 4 patients enrolled on study not available
Measure: Number; unit: Adverse Events
Arm/Group | Arm A:
Number analyzed (Participants) | 28
Adverse Events | 20

2. Secondary Outcome: Response
Description: Response rate by RECIST
Time Frame: through study completion, an average of 1 year
Population: 4 subjects did not meet physician criteria for response rate, thus their data was unusable
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A:
Number analyzed (Participants) | 28
Participants | 1

3. Secondary Outcome: To Evaluate the Secondary Endpoints of Time to Disease Progression, Duration of Response, and Overall Survival of Patients Receiving Gleevec + Temozolomide
Time Frame: through study completion
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 year
Arm/Group | Arm A:
Serious Adverse Events (participants affected / at risk) | 3/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: (N=28)
DVT (Vascular disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: (N=28)
Fatigue (General disorders) | 16 (16)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes